CLINICAL TRIAL: NCT00271960
Title: Group Prenatal Care for Reducing the Risk of STDs in Pregnant Young Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0008011972; R01MH061175 (NIH)
Record Dates: First submitted 2005-12-30; First posted 2006-01-04 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Sexually Transmitted Diseases; HIV Infections
Keywords: Pregnancy; Birth Weight; Gestational Age; Preterm Delivery; HIV Seronegativity
MeSH Terms: conditions — Sexually Transmitted Diseases; HIV Infections; Birth Weight; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Individual Care (Active Comparator): Participants will receive usual care for their prenatal visits
  Interventions: Behavioral: Usual care
- CenteringPregnancy (Active Comparator): Participants will receive CenteringPregnancy(R) group prenatal care
  Interventions: Behavioral: CenteringPregnancy
- CenteringPregnancyPlus (Experimental): Participants will receive CenteringPregancy with an HIV/STD prevention component
  Interventions: Behavioral: CenteringPregnancy; Behavioral: CenteringPregnancyPlus

INTERVENTIONS:
Behavioral: CenteringPregnancy — Following the initial intake into obstetric care in the usual manner, participants will be invited to join with 8 to 12 other women/couples/teens with similar due dates, meeting together regularly during their pregnancy.
  Arms: CenteringPregnancy; CenteringPregnancyPlus
Behavioral: CenteringPregnancyPlus — CenteringPregnancyPlus is a modified program that integrated HIV/STD prevention components with the group prenatal care model. Participants will learn skill-building in the areas of efficacy, risk assessment, negotiation skills and prevention.
  Arms: CenteringPregnancyPlus
Behavioral: Usual care — Participants will receive usual prenatal care.
  Arms: Individual Care

SUMMARY:
This study will determine the effectiveness of two group prenatal care programs as compared to individual prenatal care in reducing the risk for HIV, STDs and adverse perinatal outcomes in young women during and after pregnancy.

DETAILED DESCRIPTION:
Millions of young adults become infected with sexually transmitted diseases (STDs) each year. Young adults are particularly vulnerable to STD infection because most are not educated about STDs and use condoms improperly or inconsistently. Transmission of STDs from a pregnant woman to her baby can occur before, during, or after birth. It is, therefore, particularly important to educate young pregnant women about STDs.

Group prenatal care may be a beneficial way to assist young women. It would allow increased contact with care providers, integrate the complex needs of pregnant women, and provide support services. This study will determine the effectiveness of two group prenatal care programs as compared to individual prenatal care in reducing the risk for HIV and other STDs in young women during and after pregnancy.

Participants in this unblinded study will be randomly assigned to one of three groups: standard individual prenatal care; standard CenteringPregnancy group prenatal care; or CenteringPregnancy Plus (CP+) group prenatal care. All participants assigned to either CenteringPregnancy or CP+ will have an initial individual medical exam. Groups will be formed based on participants' estimated delivery months, and will be led by a trained independent practitioner. There will be ten 2-hour group sessions between Weeks 16 and 40 of pregnancy. At each session, participants will first weigh themselves and take their blood pressure to chart their own progress. Individual prenatal assessments lasting approximately 30 minutes will be conducted by the practitioner. Participants will then have time to fill out handouts and self-assessments and engage in discussion with other group members. Discussions will focus on education and building prenatal, childbirth, and parenting skills. The CP+ sessions will include an HIV/STD risk reduction component in addition to all the elements of the standard CenteringPregnancy program. This additional feature will consist of interactive discussion, exercises, and skill-building activities targeted towards reducing HIV/STD risk behaviors. Participants assigned to receive standard individual prenatal care will not participate in group sessions, but will receive standard prenatal care. Outcome measures will include incidence of STD infection, rapid repeat pregnancy, degree of sexual risk behavior, perinatal and psychosocial factors.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and currently at less than 24 weeks gestation
* English- or Spanish-speaking
* Willing to be randomly assigned to either group or individual prenatal care

Exclusion Criteria:

* Any severe medical problems requiring individualized assessment and tracking as a "high-risk pregnancy" (e.g., active substance use, mental illness, HIV)

Ages: 14 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1047 (Actual)
Dates: Start 2001-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Sexually transmitted disease | Measured at 2nd and 3rd trimesters and Months 6 and 12 postpartum
Rapid repeat pregnancy | Measured at Month 12 postpartum
Sexual risk behavior | Measured at 2nd and 3rd trimesters and Months 6 and 12 postpartum
Perinatal outcomes (e.g., birth weight, gestational age) | Measured at Months 6 and 12 postpartum

SECONDARY OUTCOMES:
Psychosocial factors (e.g., depression, stress, social support) | Measured at 2nd and 3rd trimesters and Months 6 and 12 postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette R. Ickovics, PhD, Principal Investigator — Yale University School of Public Health
Locations (2):
- United States (2):
  - Yale New Haven Hospital, Women's Center, New Haven, Connecticut
  - Grady Memorial Hospital, Atlanta, Georgia

REFERENCES:
- [Background] Ickovics JR. "Bundling" HIV prevention: integrating services to promote synergistic gain. Prev Med. 2008 Mar;46(3):222-5. doi: 10.1016/j.ypmed.2007.09.006. Epub 2007 Sep 29. PMID 17964637
- [Background] Massey Z, Rising SS, Ickovics J. CenteringPregnancy group prenatal care: Promoting relationship-centered care. J Obstet Gynecol Neonatal Nurs. 2006 Mar-Apr;35(2):286-94. doi: 10.1111/j.1552-6909.2006.00040.x. PMID 16620257
- [Result] Kershaw TS, Magriples U, Westdahl C, Rising SS, Ickovics J. Pregnancy as a window of opportunity for HIV prevention: effects of an HIV intervention delivered within prenatal care. Am J Public Health. 2009 Nov;99(11):2079-86. doi: 10.2105/AJPH.2008.154476. Epub 2009 Sep 17. PMID 19762662
- [Result] Ickovics JR, Kershaw TS, Westdahl C, Magriples U, Massey Z, Reynolds H, Rising SS. Group prenatal care and perinatal outcomes: a randomized controlled trial. Obstet Gynecol. 2007 Aug;110(2 Pt 1):330-9. doi: 10.1097/01.AOG.0000275284.24298.23. PMID 17666608
- [Result] Ickovics JR, Reed E, Magriples U, Westdahl C, Schindler Rising S, Kershaw TS. Effects of group prenatal care on psychosocial risk in pregnancy: results from a randomised controlled trial. Psychol Health. 2011 Feb;26(2):235-50. doi: 10.1080/08870446.2011.531577. PMID 21318932
- [Result] Gould Rothberg BE, Magriples U, Kershaw TS, Rising SS, Ickovics JR. Gestational weight gain and subsequent postpartum weight loss among young, low-income, ethnic minority women. Am J Obstet Gynecol. 2011 Jan;204(1):52.e1-11. doi: 10.1016/j.ajog.2010.08.028. Epub 2010 Oct 25. PMID 20974459
- [Result] Magriples U, Boynton MH, Kershaw TS, Duffany KO, Rising SS, Ickovics JR. Blood pressure changes during pregnancy: impact of race, body mass index, and weight gain. Am J Perinatol. 2013 May;30(5):415-24. doi: 10.1055/s-0032-1326987. Epub 2012 Oct 11. PMID 23059493
- [Result] Magriples U, Kershaw TS, Rising SS, Westdahl C, Ickovics JR. The effects of obesity and weight gain in young women on obstetric outcomes. Am J Perinatol. 2009 May;26(5):365-71. doi: 10.1055/s-0028-1110088. Epub 2008 Dec 11. PMID 19085680
- [Result] Agrawal A, Ickovics J, Lewis JB, Magriples U, Kershaw TS. Postpartum intimate partner violence and health risks among young mothers in the United States: a prospective study. Matern Child Health J. 2014 Oct;18(8):1985-92. doi: 10.1007/s10995-014-1444-9. PMID 24562504
- [Result] Cole-Lewis HJ, Kershaw TS, Earnshaw VA, Yonkers KA, Lin H, Ickovics JR. Pregnancy-specific stress, preterm birth, and gestational age among high-risk young women. Health Psychol. 2014 Sep;33(9):1033-45. doi: 10.1037/a0034586. Epub 2014 Jan 20. PMID 24447189
- [Result] Novick G, Reid AE, Lewis J, Kershaw TS, Rising SS, Ickovics JR. Group prenatal care: model fidelity and outcomes. Am J Obstet Gynecol. 2013 Aug;209(2):112.e1-6. doi: 10.1016/j.ajog.2013.03.026. Epub 2013 Mar 21. PMID 23524175
- [Result] Magriples U, Kershaw TS, Rising SS, Massey Z, Ickovics JR. Prenatal health care beyond the obstetrics service: utilization and predictors of unscheduled care. Am J Obstet Gynecol. 2008 Jan;198(1):75.e1-7. doi: 10.1016/j.ajog.2007.05.040. PMID 18166312
- [Result] Kershaw TS, Lewis J, Westdahl C, Wang YF, Rising SS, Massey Z, Ickovics J. Using clinical classification trees to identify individuals at risk of STDs during pregnancy. Perspect Sex Reprod Health. 2007 Sep;39(3):141-8. doi: 10.1363/3914107. PMID 17845525
- [Result] Westdahl C, Milan S, Magriples U, Kershaw TS, Rising SS, Ickovics JR. Social support and social conflict as predictors of prenatal depression. Obstet Gynecol. 2007 Jul;110(1):134-40. doi: 10.1097/01.AOG.0000265352.61822.1b. PMID 17601908
- [Result] Kershaw TS, Milan S, Westdahl C, Lewis J, Rising SS, Fletcher R, Ickovics J. Avoidance, anxiety, and sex: the influence of romantic attachment on HIV-risk among pregnant women. AIDS Behav. 2007 Mar;11(2):299-311. doi: 10.1007/s10461-006-9153-z. PMID 16865541
- [Derived] Kershaw TS, Arnold A, Lewis JB, Magriples U, Ickovics JR. The skinny on sexual risk: the effects of BMI on STI incidence and risk. AIDS Behav. 2011 Oct;15(7):1527-38. doi: 10.1007/s10461-010-9842-5. PMID 20976536